CLINICAL TRIAL: NCT05273697
Title: Randomized Clinical Trial to Compare Underwater Cold Snare Polypectomy (UCSP) to Conventional Cold Snare Polypectomy (CCSP) for Non Pedunculated Colon Polyps of Size 5-10mm [COLDWATER Study]
Brief Title: Clinical Study to Compare Cold Snare Underwater Polypectomy to Cold Snare Conventional Polypectomy for Colon Polyps [COLDWATER Study]
Acronym: COLDWATER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Maria Zachou, Principal Investigator, Gastroenterology Resident at Sismanogleio General Hospital, MD, MSc, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PN61759
Record Dates: First submitted 2022-02-09; First posted 2022-03-10 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Colon Polyps; Polypectomy
Keywords: colon polyps; underwater polypectomy; cold snare polypectomy; polypectomy; cold snare
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Underwater cold snare polypectomy group (Active Comparator): Cold snare polypectomy after complete immersion of the polyp in the water
  Interventions: Procedure: Underwater Cold Snare Polypectomy
- Conventional cold snare polypectomy group (Active Comparator): Cold snare polypectomy in colon lumen dilated with air
  Interventions: Procedure: Conventional Cold Snare Polypectomy

INTERVENTIONS:
Procedure: Underwater Cold Snare Polypectomy — The procedure of Underwater Cold Snare Polypectomy (UP) will be as follows:
  1. Complete suction of air from the intestinal tract
  2. Partial opening of the intestinal lumen by using sterile room temperature water via a water pump
  3. Complete immersion of the lesion in water
  4. Snaring of the lesion and a small amount of surrounding healthy tissue (1-2mm)
  5. Excision The objective will be the en bloc resection of the lesion including healthy tissue (about 2mm). If the en bloc resection fails, a piecemeal will be performed on as few specimens as possible
  Arms: Underwater cold snare polypectomy group
Procedure: Conventional Cold Snare Polypectomy — The procedure of Conventional Cold Snare Polypectomy (CCSP) will be as follows:
  1. If the entry during the endoscopy has been made with water, the water will be aspirated, and the intestinal lumen will be re-stretched using air / CO2
  2. Snaring of the lesion and a small amount of surrounding healthy tissue (1-2mm)
  3. Excision The objective will be the en bloc resection of the lesion including healthy tissue (about 2mm). If the en bloc resection fails, a piecemeal will be performed on as few specimens as possible
  Arms: Conventional cold snare polypectomy group

SUMMARY:
Colon cancer is internationally the third cause of deaths from a malignant disease. Screening colonoscopy in adults >45 years of age aims at the early diagnosis and treatment colon polyps that are precancerous lesions. Endoscopic polyp removal (polypectomy) can be done with various techniques depending on the size, morphology, location of the polyp etc. According to updated guidelines, non-pedunculated polyps of small size are treated with a cold snare in air dilated intestinal lumen (conventional cold snare polypectomy - CCSP).In recent years, several studies have described the benefits of water aided colonoscopy, as well as safety and efficacy of underwater polypectomy in large colon polyps. However, there is not enough data on small polyps which are the most commonly diagnosed.This is a prospective randomized double-blind clinical trial to compare the safety and efficacy of CCSP to underwater cold snare polypectomy (UCSP)for non-pedunculated polyps of size of 5-10 mm. A total of 398 polyps will be randomized and randomization will be performed via random numbers method of Microsoft Excel 2016. Primary outcome of this study is to determine muscularis mucosa resection rate. Secondary outcomes are the depth and percentage of R0 excisions and possible complications.

The investigators expect UCSP to ensure a higher muscularis mucosa resection rate and they attempt to examine the resection depth in the submucosal layer.These results will provide useful data for the development of guidelines in polypectomy techniques for non-pedunculated polyps 5-10mm.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 20years
2. Non pedunculated polyps (Paris classification Isp, Is, IIa, IIb)
3. Polyp size: diameter of 5 to 10mm
4. Endoscopic diagnosis of mucosal lesions - must not present malignant submucosal infiltration evidence like deepening, ulceration / ulcer, abnormal vessels, irregular surface, (NICE 1, NICE 2A, BASIC)
5. Informed consent
6. Patients who receive antiplatelet / anticoagulant therapy are included in the study only if their therapy has been modified according to ESGE guidelines

Exclusion Criteria:

1. Age <20 years old
2. Pedunculated polyps
3. Lesions with macroscopic elements of high-grade dysplasia or submucosal infiltration
4. Sites with previous polypectomy
5. Patients with idiopathic inflammatory bowel disease
6. Patients with coagulation disorders
7. Patients with severe organ failure

7.Patients who during endoscopy will undergo any technique using electrocautery / electrocoagulation will not be eligible for participation in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-06-11 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
percentage of muscularis mucosa included in specimen (%) | through study completion, an average of 1 year
  Determination of percentage of muscularis mucosa included in specimen. The determination of the percentage of the area containing muscularis mucosa layer will be done by measuring the length of muscularis mucosa mm / length of specimen mm x100%. Using an ocular and stage micrometer, the length of the muscularis mucosa underlining a neoplastic lesion was measured, along with the specimen's maximum diameter (mm)

SECONDARY OUTCOMES:
Presence or absence of submucosal in the specimen and its depth (if present) | through study completion, an average of 1 year
  Presence or absence of submucosa
  - Measurement of submucosa depth in μm (when submucosa is present in the specimen)
Percentage of R0 Resections | through study completion, an average of 1 year
  Vial 1 : Determination of polypectomy margin according to Residual Tumor Classification Vial 1A : Determination of horizontal margins: presence of residual damage or not In order to determine the horizontal margins, 2-4 biopsies will be taken from the resection area (2 biopsies antidiametrically in polyps of 5-7 mm size, 4 biopsies in polyps of 8-10 mm size). One cup of forceps will be placed in the defect and the second in the macroscopically normal mucosa.
  The received tissue pieces will be placed in a new vial with formol (Vial 1A)
  A microscopically margin-negative resection will be characterized as "R0 resection" The determination of R0 Resection Rate will be done by measuring the number of R0 resections / number of all the resections regardless R classification
Complication rate | 30 days after the polypectomy (treatment procedure)
  intraprocedural bleeding, post-procedural bleeding, perforation, abdominal pain not due to perforation. These complications will be evaluated by a study physician of the Gastroenterology Department with a phone call and clinical examination if needed
Recurrence lesion rate during repeat colonoscopy in 6-12months | 6-12 months after polypectomy (treatment procedure)
  A subgroup of the sample size will undergo a follow up colonoscopy in 6-12 months in order to identify lesion recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Maria Zachou, MD,Msc, Principal Investigator — Department of Gastroenterology, General Hospital of Athens Sismanogleio, Greece; Stylianos Kykalos, Assist.Prof, Study Director — 2nd Department of Propaedeutic Surgery, National and Kapodistrian University of Athens, General Hospital Laiko, Athens, Greece; Evangelos Kalaitzakis, Assist.Prof, Study Chair — Department of Gastroenterology, University Hospital of Heraklion, University of Crete, Heraklion, Greece; Stavros Sougioultzis, Study Chair — Gastroenterology Unit, Department of Pathophysiology, School of Medicine, National and Kapodistrian University Athens, Greece
Locations (1):
- Sismanogleio General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
Available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Zachou M, Varytimiadis K, Androutsakos T, Katsaras G, Zoumpouli C, Lalla E, Nifora M, Karantanos P, Nikiteas N, Sougioultzis S, Kalaitzakis E, Kykalos S. Protocol design for randomized clinical trial to compare underwater cold snare polypectomy to conventional cold snare polypectomy for non-pedunculated colon polyps of size 5-10 mm (COLDWATER study). Tech Coloproctol. 2023 Apr;27(4):325-333. doi: 10.1007/s10151-022-02731-9. Epub 2022 Nov 18. PMID 36399201

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT05273697/Prot_SAP_000.pdf